CLINICAL TRIAL: NCT04963907
Title: Randomised Controlled Trial of the Clinical and Cost Effectiveness of Alpha-Stim AID Cranial Electrotherapy Stimulation (CES) in Treatment Seeking Patients With Moderate Severity Depressive Episodes in Primary Care
Brief Title: Alpha-Stim AID and Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Electromedical Products International, Inc. (Industry)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UK-MDDNHS
Record Dates: First submitted 2021-06-25; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Alpha-Stim; Cranial Electrotherapy Stimulation (CES)
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: The study is a multi-centre parallel group, double blind, non-commercial, randomised controlled trial (RCT).
Who Masked: Participant, Investigator
Masking Description: Devices are programmed by the manufacturer prior to shipping to investigator. Active devices are programmed at 100 uA for 60 minutes, which is subsensory. Sham devices will display 100 uA and count down from 60 minutes, but will not emit a current. Neither the investigators nor the participants will know which devices are active and which are sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active CES Therapy (Active Comparator): Participants will be asked to use Alpha-Stim 60 minutes daily for 8 weeks. Active devices are programmed to emit a current intensity of 100 uA at 0.5 Hz and will be programmed to run for 60 minutes. Participants will not be able to adjust the settings on the devices.
  Interventions: Device: Active Alpha-Stim CES
- Sham CES Therapy (Sham Comparator): Participants will be asked to use Alpha-Stim 60 minutes daily for 8 weeks. Sham devices are programmed to display a current intensity of 100 uA at 0.5 Hz and will be programmed to run for 60 minutes, but no current will be emitted from the device. Participants will not be able to adjust the settings on the devices.
  Interventions: Device: Sham Alpha-Stim CES

INTERVENTIONS:
Device: Active Alpha-Stim CES — Active Alpha-Stim devices will be randomly assigned to participants for use daily for 8 weeks.
  Arms: Active CES Therapy
Device: Sham Alpha-Stim CES — Sham Alpha-Stim devices will be randomly assigned to participants for use daily for 8 weeks.
  Arms: Sham CES Therapy

SUMMARY:
The study will be a multi-centre parallel group, double blind, non-commercial, randomised controlled superiority trial. Study participants will be referred from Primary Care GP practices via their GP and randomised into active Alpha-Stim AID Cranial Electrotherapy Stimulations (CES) or sham Alpha-Stim AID CES.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years and above. There is no maximum age limit.
* Diagnosis of current Major Depressive Episode (MDE). This will be confirmed using the research version of the Structured Clinical Interview for DSM-5 (SCID-5-RV) at baseline.
* A Score of ≥10 to 19 on 9-item self-rated Personal Health Questionnaire (PHQ-9).
* Have either been offered the option of antidepressant medication or have been prescribed antidepressant medication for a minimum of 6 weeks in the last 3 months.
* Capable of giving oral and written informed consent to the study.
* Agrees to return Alpha-Stim equipment at the end of the study and not to purchase this equipment privately during the study.

Exclusion Criteria:

* A score of ≥20 on the PHQ-9.
* Neurological conditions e.g. brain neoplasm, cerebrovascular events, epilepsy, neurodegenerative disorders, and prior brain surgery
* Requires urgent clinical care such as having persistent suicidal ideation, self-harm or suicidal intent.
* Known to be pregnant.
* Implantation with a pace maker, cochlear implant or an implantable cardioverter device (ICD).
* Major unstable medical illness requiring further investigation or treatment.
* A diagnosis of current substance use disorder or dependence, dementia, eating disorder, bipolar disorder or non-affective psychosis because the use of CES treatment would otherwise require additional supervision or is associated with additional risk e.g. of mania in bipolar disorder. Determination of these conditions will be confirmed using a diagnostic clinical interview (SCID-5-RV).
* Completed and benefitted from/responded to psychological treatment for depression in the last 3 months or planning to commence psychological treatment in the next 6 months.
* Involved with any other clinical trial at the time of consent or 6 months prior.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in depression | 16 weeks
  Determine if there is a significant difference from baseline to 16 weeks on the Grid version of the Hamilton Depression Scale. The GRID-HAMD is a 17 item scale with scores ranging from 0-54. Higher scores indicate increased severity of depression. Scores of 0-7 is generally accepted to be within the normal range (clinical remission) and a score of 20 or above indicates moderate severity.

SECONDARY OUTCOMES:
Cost effectiveness | 16 weeks
  This will be analysed through the measurement of costs from personal, health and social care perspectives using Client Service Receipt inventory at 4, 8 and 16 weeks. The CSRI is a measure of the full health and social care cost and patient cost of treatment.
Change in anxiety | 16 weeks
  Determine if there is a significant difference from baseline to 16 weeks on the Generalized Anxiety Disorder Scale. The GAD-7 is a 7-item self-rated measure of the severity of Generalized Anxiety Disorder. Scores range from 0-21. Scores of 5, 10, 15 and 20 represent cut off points for mild, moderate, moderately severe and severe anxiety.
Change in quality of life - work and social functioning | 16 weeks
  Determine if there is a significant difference in quality of life related to work and social functioning from baseline to 16 weeks, as measured by the Work and Social Adjustment Scale. The WASA is a 5-item self-rated measure of work and social function. The maximum score of the WSAS is 40, lower scores indicate less impairment in functioning.
Change in quality of life - health related | 16 weeks
  Determine if there is a significant difference in quality of life related to overall health using a standardized measure developed by the Euroqual group. EQ5D-5L is 5 item standardized instrument for measuring generic health status. It is used by NICE to generate quality adjusted life years for cost effectiveness assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Morriss, MD, Principal Investigator — University of Nottingham Research and Innovation
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No